CLINICAL TRIAL: NCT04202718
Title: VitalConnect VitalPatch ECG Interpretation/Arrhythmia Detection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started due to COVID-19 pandemic
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Ashok Palagiri, Physician, Mercy Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-007
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Arrythmia, Cardiac
Keywords: ECG Interpretation
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single group (Other): Where a wearable biosensor is being considered for use in the health management of individuals at high-risk for poor health outcomes, and in the detection or prevention of adverse events within settings where traditional monitoring devices are not currently in use, the ECG interpretation will provide Arrhythmia detection which will help ensure that irregular rhythms will be reported quickly.
  Interventions: Diagnostic Test: VitalPatch Device

INTERVENTIONS:
Diagnostic Test: VitalPatch Device — The VitalPatch® is an IRB (791130) and FDA approved wearable device that allows for the constant monitoring of biometric measurements and may have utility in the health management of individuals at high-risk for poor health outcomes and in the detection or prevention of adverse events within settings where more traditional telemetry monitoring devices are not currently in use.

SUMMARY:
Subjects in this study will wear the VitalPatch with the added ECG Interpretation and arrhythmia detection features which will expedite the identification of patients whose condition may rapidly deteriorate as well as eliminate the majority of non-actionable alarms.

DETAILED DESCRIPTION:
This project intends to validate, through comparative study, the output of new technologies (ECG Interpretation and arrhythmia detection) to the VistaCenter platform, aiming to replace current telemetry monitoring equipment. The new technology, through the previous Mercy pilot study, has demonstrated greater accuracy in the detection of ventricular tachycardia patterns and other dysrhythmias/arrhythmias, as well as, reducing the volume of false alarms resulting in the mitigation of alarm fatigue experienced by bedside staff and monitor technicians.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* No skin trauma to the site where the patch will be applied
* No known allergies to hydrocolloid or silicone based adhesives
* Admitted to Mercy Hospital Washington Cardiac Unit on the 5th floor and have been placed in one of the assigned rooms and require cardiac/telemetry monitoring as ordered by their physician

Exclusion Criteria:

* Pacemaker or Implanted Defibrillator (ICD)
* Pregnancy
* Adults unable to provide informed consent
* Individuals who cannot read and understand English
* Prisoners
* Not recommended for use in MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in false alarms received from current telemetry monitoring technology | 6 months
  • Compare generation of false alarms with VitalPatch and current telemetry monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Hospital Washington, Washington, Missouri, United States